CLINICAL TRIAL: NCT00037466
Title: Relation of Diet to Serum Homocysteine Level in Youths
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Voula Osganian, Associate Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: 1173; R01HL066643 (NIH)
Record Dates: First submitted 2002-05-16; First posted 2002-05-17 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2005-02

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To examine the relation between diet and plasma total homocysteine levels in an ethnically and geographically diverse cohort of adolescents.

DETAILED DESCRIPTION:
BACKGROUND:

Data from observational studies suggest that plasma total homocysteine (tHcy) concentration may be an independent and modifiable risk factor for cardiovascular disease (CVD) in adults. Plasma tHcy levels respond rapidly to nutrient supplementation with folic acid and vitamins Bl2 and B6, alone or in combination. The available data and the potential for prevention provide a strong rationale for understanding determinants of tHcy in youth. However, no large U.S. studies have examined the relation between tHcy levels to individuals' dietary intakes of folic acid and vitamins Bl2 and B6 in youth.

DESIGN NARRATIVE:

During the Child and Adolescent Trial for Cardiovascular Health (CATCH) Phase 3, a cross-sectional study of serum tHcy levels was conducted in eighth grade students (Jan-June 1997). Higher mean levels of plasma total homocysteine were observed among males, Blacks, and non-users of multi-vitamins and a strong, inverse association with serum levels of folic acid and to a lesser extent, with serum vitamin Bl2. A second measurement of the cohort at grade 12 was conducted in order to assess the dose-response relation between serum tHcy and dietary intakes (not measured in grade 8) of folic acid, vitamin B12 and vitamin B6. In addition and of equal importance, changes were evaluated in serum folic acid and tHcy levels from grade 8 to 12, after full implementation of fortification of cereal and grain products in the U.S. with folic acid and its impact on the distribution of tHcy levels in adolescents described. Effective January 1, 1998, the U.S. Department of Agriculture mandated the addition of folic acid to all flour and grain products in the United States. CATCH had a unique opportunity to examine the effect of "this natural experiment" on the distribution of serum tHcy in the cohort, because serum tHcy levels were measured in grade 8, just prior to full implementation of the mandate. Furthermore, the study had adequate sample size to examine these changes among important demographic subgroups such as, males vs. females and Caucasians vs. African Americans vs. Hispanics. Information generated by this study will be valuable for designing specific dietary interventions for youth and targeting subgroups of children who may be at higher risk for CVD.

ELIGIBILITY:
The subjects for this analysis were had to be part of CATCH, a trial designed to evaluate the effectiveness of a multi-component school-based cardiovascular health promotion intervention, described elsewhere in detail(29-30). The main trial (1991-1994) was conducted among students in grades 3-5 attending 96 public elementary schools (56 intervention and 40 control schools) in California, Louisiana, Minnesota, and Texas. Following the main trial, two observational studies were conducted that measured physiologic and behavioral risk factors in study participants from grades 6 to 8 (1994-1997) (pre-fortification) and in grade 12 (post-fortification) (2000-2001).

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The CATCH study initially recruited 5,106 third grade students to participate in a risk factor screening at baseline. Of these, 3645 (71%) participated in risk factor screening at the end of grade 8 when serum tHcy, folate, vitamin B6 and vitamin B12 were first assessed and 2909 (57%) students participated in the follow-up risk factor screening in grade 12. Of these students, 2445, attended both grade 8 and grade 12 examinations and provided blood at both examinations. This group constituted the study population for this report.
Sampling Method: Non-Probability Sample
Enrollment: 2445 (Actual)
Dates: Start 2000-09; Primary Completion 2001-08 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Serum homocysteine (tHcy) concentrations | 4 years
Serum folic acid concentrations | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Stavroula Osganian, MD, ScD, Principal Investigator — Boston Children's Hospital

IPD SHARING:
Plan to Share IPD: No
Data Sharing was not required at the time the study was conducted.

REFERENCES:
- [Result] Enquobahrie DA, Feldman HA, Hoelscher DH, Steffen LM, Webber LS, Zive MM, Rimm EB, Stampfer MJ, Osganian SK. Serum homocysteine and folate concentrations among a US cohort of adolescents before and after folic acid fortification. Public Health Nutr. 2012 Oct;15(10):1818-26. doi: 10.1017/S1368980012002984. PMID 22974678
- See also: Final Results Paper — http://www.ncbi.nlm.nih.gov/pubmed/22974678